CLINICAL TRIAL: NCT01288495
Title: Investigation of Supplemental L-alanine in the Management of Dietary Fructose Intolerance: a Double-blind, Randomized Crossover Study
Brief Title: Randomized Control Trial of L-Alanine and Placebo in Fructose Intolerance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI moved institutions and changed study protocol
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Satish Rao, PI, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Long Term Fructose
Record Dates: First submitted 2011-01-31; First posted 2011-02-02 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Dietary Fructose Intolerance
MeSH Terms: interventions — Psyllium

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- L-alanine (Experimental): Subjects will consume l-alanine prior to eating fructose-containing foods.
  Interventions: Dietary Supplement: supplemental L-alanine
- Placebo (Placebo Comparator): Subjects will consume the placebo prior to eating fructose-containing foods.
  Interventions: Dietary Supplement: Metamucil

INTERVENTIONS:
Dietary Supplement: supplemental L-alanine — Subjects will consume l-alanine prior to eating fructose-containing foods.
  Arms: L-alanine
Dietary Supplement: Metamucil — Subjects will consume the placebo prior to eating fructose-containing foods.
  Arms: Placebo

SUMMARY:
Data suggest that alanine may facilitate the intestinal absorption of fructose in patients with DFI and thereby may decrease GI symptoms.

We hypothesize that the ingestion of supplemental L-alanine along with mixed meals or snacks that contain foods with free fructose or high fructose content will decrease GI symptoms in subjects with dietary fructose intolerance by facilitating intestinal absorption of fructose.

Aim: To investigate the effects of co- administration of equi-molar doses of L-alanine or placebo on the occurrence of GI symptoms in subjects with dietary fructose intolerance, in a randomized, double blind, cross over study.

Methods: We propose to investigate the effects of co-administration of equi-molar doses of L-alanine or placebo on the occurrence of GI symptoms in 70 subjects with dietary fructose intolerance, in a randomized, double blind, cross over study.

Data Analysis: The primary outcome measure will be a comparison of baseline breath sample values and study visit breath sample values. Additionally, we will assess subject-reported occurence and severity of nine gastrointestinal symptoms during the test on a visual analog scale (VAS).

Expected Results: We anticipate that dietary fructose intolerance (DFI) symptoms will improve with ingestion of supplemental L-alanine (along with foods containing free fructose or high fructose content). We additionally expect treatment of DFI with administration of L-alanine powder to be more practical than co-ingestion of alanine-rich foods, and more convenient for patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-99 years
2. Diagnosis of fructose malabsorption (positive breath test after ingestion of 25 grams of fructose defined as either (a) ≥ 20 ppm rise of breath H2/CH4/both over baseline values or a successive rise of ≥ 5 ppm over baseline and in 3 consecutive breath samples)

Exclusion Criteria:

1. Cognitive impairment or any other inability to provide informed consent
2. Prisoners
3. GI surgery except appendectomy, cholecystectomy, caesarean section, hysterectomy
4. Antibiotics in the previous 6 weeks
5. History of bacterial overgrowth or lactose intolerance
6. Major co-morbid illnesses, including chronic pancreatitis, celiac disease, inflammatory bowel disease, diabetes, scleroderma, pseudo-obstruction syndromes etc.
7. Known food allergies
8. Medication use: opioids, Tegaserod, laxatives, enemas
9. An allergy or intolerance to any fiber supplements or other dietary nutritional supplements such as: psyllium (Metamucil), Maltodextrin, Citric Acid, and methylcellulose (Citrucel).
10. Difficulty swallowing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
GI symptom score | 4 weeks
  Change in GI symptom score with alanine & placebo, when compared to the baseline

SECONDARY OUTCOMES:
Fructose consumption | 4 weeks
  Estimated daily consumption of fructose during the alanine & placebo phases, when compared to baseline using prospective food diaries
Breath hydrogen and methane | 4 weeks
  Changes in Breath hydrogen and/or methane values with Alanine and Placebo when compared with baseline
Quality of life (SF-12) | 4 weeks
  Changes in SF-12 scores between baseline and after alanine and placebo

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States